CLINICAL TRIAL: NCT01689363
Title: A Randomized, Double-Blinded, Negative- and Positive-Controlled Study for Evaluation of the Allergenicity of Amphadase® in Healthy Volunteers Using Intradermal Skin Test
Brief Title: Evaluation of the Allergenicity of AMPHADASE INJECTION (Hyaluronidase Injection USP)
Acronym: H001-A2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: API-H001-CLN-A2
Record Dates: First submitted 2012-09-13; First posted 2012-09-21 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Allergic Skin Reaction
Keywords: hyaluronidase; enzymes with tissue spreading activity; allergic reaction; intradermal skin testing
MeSH Terms: conditions — Hypersensitivity | interventions — Hyaluronoglucosaminidase; Chondroitinases and Chondroitin Lyases; Histamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm H (Experimental): Intradermal injection of Amphadase (hyaluronidase 150 USP units/mL)
  Interventions: Drug: Hyaluronidase
- Arm P (Active Comparator): Intradermal injection of Histatrol (histamine base 0.1 mg/mL)
  Interventions: Drug: Histamine
- Arm N (Placebo Comparator): Intradermal injection of saline (0.02 mL)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Hyaluronidase — Subjects received intradermal injections of 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at two random sites on their forearms.
  Other Names: Amphadase®
  Arms: Arm H
Drug: Histamine — Subjects received one intradermal injection of 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at one random sites on their forearms.
  Other Names: Histatrol®
  Arms: Arm P
Drug: Saline — Subjects received one intradermal injection of 0.02 mL saline at one random site on their forearm.
  Arms: Arm N

SUMMARY:
This study is designed to evaluate the allergenicity of Amphadase® in healthy volunteers using an intradermal skin test.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers of either gender; Those without clinically significant cardiovascular gastrointestinal, hepatic, neurological, psychiatric, endocrine, or other major systemic disease that would unduly risk the subject's safety or interfere with the interpretation of results, assessed according to the judgment of the Principal Investigator. A non-inclusive list which would not be exclusionary and define healthy individual for the purposes of this study are:

* hypothyroidism,
* stable hypertension except those subjects on beta blockers including ocular preparations,
* seasonal/perennial allergic rhinitis if able to wash out of antihistamines,
* stable, mild intermittent asthma (subjects using beta agonists as a monotherapy on an as-needed basis, excluding daily usage),
* migraine if not taking excluded medications,
* mild anxiety/depression if not taking excluded medications, and
* mild arthritic conditions if not taking excluded medications.

  * Willingness and ability to sign an informed consent document;
  * 18 - 80 years of age;
  * Intact skin at the forearm ;
  * Female participants are currently practicing effective birth control methods or abstinence.

Exclusion Criteria:

* Known allergy, hypersensitivity or contraindications to hyaluronidase, thimerosal, edetate disodium (EDTA);
* Use of medications within a duration considered to interfere with skin testing.
* Known dermographism which may interfere with skin testing.
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selina Su, MPH, Study Chair — A:mphastar Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Amphastar Site 0022, Eugene, Oregon
  - Amphastar Site 0023, Lake Oswego, Oregon
  - Amphastar Site 0026, Portland, Oregon
  - Amphastar Site 0038, Renton, Washington
  - Amphastar Site 0034, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barr J, Kirkpatrick N, Dick A, Leonard L, Hawksworth G, Noble DW. Effects of adrenaline and hyaluronidase on plasma concentrations of lignocaine and bupivacaine after peribulbar anaesthesia. Br J Anaesth. 1995 Dec;75(6):692-7. doi: 10.1093/bja/75.6.692. PMID 8672315
- [Background] Brydon CW, Basler M, Kerr WJ. An evaluation of two concentrations of hyaluronidase for supplementation of peribulbar anaesthesia. Anaesthesia. 1995 Nov;50(11):998-1000. doi: 10.1111/j.1365-2044.1995.tb05940.x. PMID 8678264
- [Background] Ahluwalia HS, Lukaris A, Lane CM. Delayed allergic reaction to hyaluronidase: a rare sequel to cataract surgery. Eye (Lond). 2003 Mar;17(2):263-6. doi: 10.1038/sj.eye.6700243. No abstract available. PMID 12640426
- [Background] Agrawal A, McLure HA, Dabbs TR. Allergic reaction to hyaluronidase after a peribulbar injection. Anaesthesia. 2003 May;58(5):493-4. doi: 10.1046/j.1365-2044.2003.03154_17.x. No abstract available. PMID 12694021
- [Background] Kempeneers A, Dralands L, Ceuppens J. Hyaluronidase induced orbital pseudotumor as complication of retrobulbar anesthesia. Bull Soc Belge Ophtalmol. 1992;243:159-66. PMID 1302146
- [Background] Minning CA Jr. Hyaluronidase allergy simulating expulsive choroidal hemorrhage. Arch Ophthalmol. 1994 May;112(5):585-6. doi: 10.1001/archopht.1994.01090170029012. No abstract available. PMID 8185511
- [Background] Szepfalusi Z, Nentwich I, Dobner M, Pillwein K, Urbanek R. IgE-mediated allergic reaction to hyaluronidase in paediatric oncological patients. Eur J Pediatr. 1997 Mar;156(3):199-203. doi: 10.1007/s004310050582. PMID 9083759
- [Background] Allergy testing. American College of Physicians. Ann Intern Med. 1989 Feb 15;110(4):317-20. No abstract available. PMID 2578014
- [Background] Poulsen LK. In vivo and in vitro techniques to determine the biological activity of food allergens. J Chromatogr B Biomed Sci Appl. 2001 May 25;756(1-2):41-55. doi: 10.1016/s0378-4347(01)00070-6. PMID 11419727
- [Background] Howard A, Mercer P, Nataraj HC, Kang BC. Bevel-down superior to bevel-up in intradermal skin testing. Ann Allergy Asthma Immunol. 1997 Jun;78(6):594-6. doi: 10.1016/s1081-1206(10)63222-x. PMID 9207725
- [Background] Barbaud A, Reichert-Penetrat S, Trechot P, Jacquin-Petit MA, Ehlinger A, Noirez V, Faure GC, Schmutz JL, Bene MC. The use of skin testing in the investigation of cutaneous adverse drug reactions. Br J Dermatol. 1998 Jul;139(1):49-58. doi: 10.1046/j.1365-2133.1998.02313.x. PMID 9764148
- [Background] Fisher MM, Bowey CJ. Intradermal compared with prick testing in the diagnosis of anaesthetic allergy. Br J Anaesth. 1997 Jul;79(1):59-63. doi: 10.1093/bja/79.1.59. PMID 9301390
- [Background] Ruzicka T, Gerstmeier M, Przybilla B, Ring J. Allergy to local anesthetics: comparison of patch test with prick and intradermal test results. J Am Acad Dermatol. 1987 Jun;16(6):1202-8. doi: 10.1016/s0190-9622(87)70158-3. PMID 3597862

RESULTS

PARTICIPANT FLOW:
Groups:
- H, N, H, P: Subjects received four intradermal injections where study drug was injected to sites on the subject's forearms in the following order: 1) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the upper-left forearm; 2) 0.02 mL saline at the lower-left forearm; 3) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the upper-right forearm; 4) 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at the lower-right forearm
- H, N, P, H: Subjects received four intradermal injections where study drug was injected to sites on the subject's forearms in the following order: 1) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the upper-left forearm; 2) 0.02 mL saline at the lower-left forearm; 3) 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at the upper-right forearm; 4) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the lower-right forearm
- H, P, H, N: Subjects received four intradermal injections where study drug was injected to sites on the subject's forearms in the following order: 1) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the upper-left forearm; 2) 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at the lower-left forearm; 3) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the upper-right forearm; 4) 0.02 mL saline at the lower-right forearm
- H, P, N, H: Subjects received four intradermal injections where study drug was injected to sites on the subject's forearms in the following order: 1) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the upper-left forearm; 2) 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at the lower-left forearm; 3) 0.02 mL saline at the upper-right forearm; 4) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the lower-right forearm
- N, H, H, P: Subjects received four intradermal injections where study drug was injected to sites on the subject's forearms in the following order: 1) 0.02 mL saline at the upper-left forearm; 2) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the lower-left forearm; 3) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the upper-right forearm; 4) 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at the lower-right forearm
- N, H, P, H: Subjects received four intradermal injections where study drug was injected to sites on the subject's forearms in the following order: 1) 0.02 mL saline at the upper-left forearm; 2) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the lower-left forearm; 3) 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at the upper-right forearm; 4) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the lower-right forearm
- P, H, H, N: Subjects received four intradermal injections where study drug was injected to sites on the subject's forearms in the following order: 1) 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at the upper-left forearm; 2) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the lower-left forearm; 3) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the upper-right forearm; 4) 0.02 mL saline at the lower-right forearm
- P, H, N, H: Subjects received four intradermal injections where study drug was injected to sites on the subject's forearms in the following order: 1) 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at the upper-left forearm; 2) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the lower-left forearm; 3) 0.02 mL saline at the upper-right forearm; 4) 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at the lower-right forearm
Period: Overall Study
Arm/Group | H, N, H, P | H, N, P, H | H, P, H, N | H, P, N, H | N, H, H, P | N, H, P, H | P, H, H, N | P, H, N, H
Started | 32 | 32 | 32 | 31 | 31 | 31 | 32 | 32
Completed | 32 | 31 | 32 | 31 | 31 | 31 | 32 | 32
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Study Population: Subjects received four intradermal injections of study drug (two injections of 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL), one injection of 0.02 mL Histatrol® (histamine base 0.1 mg/mL), one injection of 0.02 mL saline) in a random order at four locations on the subjects' forearms.
Arm/Group | Total Study Population
Number analyzed (Participants) | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 239
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 126
Region of Enrollment [Number; unit: participants]
  United States | 253

OUTCOME MEASURES:

1. Primary Outcome: Positive Allergic Reaction to Amphadase® in the Per-Protocol Population (PPP)
Description: Subjects received intradermal injections at 4 injection sites following a randomized configuration of study medications. Injection sites were monitored for any characteristic immediate reactions after the study drug injections. A positive reaction consisted of: a) reaction appearing within 30 minutes of drug placement; b) wheal (>8 mm) with or without pseudopods; c) reaction accompanying erythema; and d) reaction accompanying localized itching.
Time Frame: Up to 30 minutes after the final study drug injection
Population: Subjects who: a) have received the right treatment; b) have a negative reaction for the negative control; c) have a positive reaction for the positive control; and d) have the same reaction for both Amphadase® treatments
Measure: Number; unit: participants
Groups:
- Per-Protocol Population (PPP): Subjects who: a) have received the right treatment; b) have a negative reaction for the negative control; c) have a positive reaction for the positive control; and d) have the same reaction for both Amphadase® treatments
Arm/Group | Per-Protocol Population (PPP)
Number analyzed (Participants) | 183
participants | 0

2. Primary Outcome: Positive Allergic Reaction to Amphadase® in the Intent-to-Treat Population (ITT)
Description: as for outcome 1
Time Frame: Up to 30 minutes after the final study drug injection
Population: Subjects who have been randomized
Measure: Number; unit: participants
Groups:
- Intent-to-Treat Population (ITT): Subjects who have been randomized
Arm/Group | Intent-to-Treat Population (ITT)
Number analyzed (Participants) | 253
participants | 7

3. Secondary Outcome: Observed Wheal Size in the Per-Protocol Population (PPP)
Description: Subjects received intradermal injections at 4 injection sites following a randomized configuration of study medications. Injection sites were monitored for any characteristic immediate reactions after the study drug injections. The observed wheal size is the greatest wheal diameter measured at the injection site(s) for a specific study drug injection.
Time Frame: Up to 30 minutes after the final study drug injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Arm H: Subjects received intradermal injections of 0.02 mL Amphadase® (hyaluronidase 150 USP units/mL) at two sites on their forearms
- Arm N: Subjects received an intradermal injection of 0.02 mL saline at one site on their forearms
- Arm P: Subjects received an intradermal injection of 0.02 mL Histatrol® (histamine base 0.1 mg/mL) at one site on their forearms
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 183 | 183 | 183
mm | 1.1 (2.6) | 1.7 (2.7) | 15.3 (4.9)

4. Secondary Outcome: Observed Erythema Size in the Per-Protocol Population (PPP)
Description: Subjects received intradermal injections at 4 injection sites following a randomized configuration of study medications. Injection sites were monitored for any characteristic immediate reactions after the study drug injections. The observed erythema size is the greatest erythema diameter measured at the injection site(s) for a specific study drug injection.
Time Frame: Up to 30 minutes after the final study drug injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 183 | 183 | 183
mm | 4.3 (7.0) | 0.6 (3.7) | 44.4 (11.7)

5. Secondary Outcome: Allergic Wheal Size in the Per-Protocol Population (PPP)
Description: Subjects received intradermal injections at 4 injection sites following a randomized configuration of study medications. Injection sites were monitored for any characteristic immediate reactions after the study drug injections. The allergic wheal size is the greatest wheal diameter with accompanying erythema and localized itching measured at the injection site(s) for a specific study drug injection.
Time Frame: Up to 30 minutes after the final study drug injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 183 | 183 | 183
mm | 0.1 (0.9) | 0.0 (0.0) | 15.2 (4.9)

6. Secondary Outcome: Allergic Erythema Size in the Per-Protocol Population (PPP)
Description: Subjects received intradermal injections at 4 injection sites following a randomized configuration of study medications. Injection sites were monitored for any characteristic immediate reactions after the study drug injections. The allergic erythema size is the greatest erythema diameter with accompanying localized itching measured at the injection site(s) for a specific study drug injection.
Time Frame: Up to 30 minutes after the final study drug injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 183 | 183 | 183
mm | 1.1 (5.0) | 0.0 (0.1) | 44.1 (11.8)

7. Secondary Outcome: Local Itchiness Rate in the Per-Protocol Population (PPP)
Description: Subjects received intradermal injections at 4 injection sites following a randomized configuration of study medications. Injection sites were monitored for any characteristic immediate reactions after the study drug injections. The local itchiness rate is the percentage of subjects that reported localized itching at the injection site(s) for a specific study drug injection.
Time Frame: Up to 30 minutes after the final study drug injection
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 183 | 183 | 183
percentage of participants | 7.7 | 1.1 | 100.0

8. Secondary Outcome: Erythema Responder Rate in the Per-Protocol Population (PPP)
Description: Subjects received intradermal injections at 4 injection sites following a randomized configuration of study medications. Injection sites were monitored for any characteristic immediate reactions after the study drug injections. The erythema responder rate is the percentage of subjects that showed an erythema reaction at the injection site(s) for a specific study drug injection.
Time Frame: Up to 30 minutes after the final study drug injection
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 183 | 183 | 183
percentage of participants | 51.4 | 8.7 | 100.0

9. Secondary Outcome: Observed Wheal Size in the Intent-to-Treat Population (ITT)
Description: as for outcome 3
Time Frame: Up to 30 minutes after the final study drug injection
Population: Subjects who have been randomized
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 253 | 253 | 253
mm | 1.5 (3.3) | 1.7 (2.8) | 14.1 (5.6)

10. Secondary Outcome: Observed Erythema Size in the Intent-to-Treat Population (ITT)
Description: as for outcome 4
Time Frame: Up to 30 minutes after the final study drug injection
Population: Subjects who have been randomized
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 253 | 253 | 253
mm | 5.4 (9.6) | 0.9 (4.5) | 41.5 (14.7)

11. Secondary Outcome: Allergic Erythema Size in the Intent-to-Treat Population (ITT)
Description: as for outcome 6
Time Frame: Up to 30 minutes after the final study drug injection
Population: Subjects who have been randomized
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 253 | 253 | 253
mm | 2.1 (8.0) | 0.1 (1.9) | 34.0 (21.1)

12. Secondary Outcome: Local Itchiness Rate in the Intent-to-Treat Population (ITT)
Description: as for outcome 7
Time Frame: Up to 30 minutes after the final study drug injection
Population: Subjects who have been randomized
Measure: Number; unit: percentage of participants
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 253 | 253 | 253
percentage of participants | 10.3 | 1.6 | 79.1

13. Secondary Outcome: Erythema Responder Rate in the Intent-to-Treat Population (ITT)
Description: as for outcome 8
Time Frame: Up to 30 minutes after the final study drug injection
Population: Subjects who have been randomized
Measure: Number; unit: percentage of participants
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 253 | 253 | 253
percentage of participants | 53.8 | 11.1 | 97.6

14. Secondary Outcome: Allergic Wheal Size in the Intent-to-Treat Population (ITT)
Description: as for outcome 5
Time Frame: Up to 30 minutes after the final study drug injection
Population: Subjects who have been randomized
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm H | Arm N | Arm P
Number analyzed (Participants) | 253 | 253 | 253
mm | 0.5 (2.4) | 0.0 (0.7) | 11.5 (7.6)

ADVERSE EVENTS:
Time Frame: Signing of Informed Consent until Adverse Event Resolution/Stabilization (approximately 30 days)
Description: Adverse drug events (ADEs), whether observed by investigators or reported by the subjects, will be documented, evaluated, followed up, and treated if deemed necessary. ADEs will be followed until stabilized/resolved or 30 days from the date the subject has finished the study, whichever is sooner.
Groups:
- All Arms: Cannot identify which study drug may be associated with the ADE because the subject received all four injections almost at the same time
Arm/Group | Arm H | Arm N | Arm P | All Arms
Serious Adverse Events (participants affected / at risk) | 0/253 | 0/253 | 0/253 | 0/253
Other Adverse Events (participants affected / at risk) | 0/253 | 0/253 | 0/253 | 0/253

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other